CLINICAL TRIAL: NCT07224542
Title: Smart Soft Contact Lenses for Continuous 24-hour Monitoring of Intraocular Pressure in Glaucoma Care
Brief Title: Smart Soft Contact Lenses for Monitoring Glaucoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Eye Institute (NEI) (NIH); Purdue University (Other)
Responsible Party: Principal Investigator, Pete Kollbaum, OD, PhD, Associate Dean, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IU-24139; R01EY034901 (NIH)
Record Dates: First submitted 2025-10-17; First posted 2025-11-04 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
Keywords: glaucoma; contact lens; sensor; eye pressure; IOP; optometry; ophthalmology
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Sensor Experimental Arm (Experimental): Followed with device and comparator
  Interventions: Device: Bare Contact Lens; Device: Clinical IOP Measure; Device: Experimental Contact Lens Sensor

INTERVENTIONS:
Device: Bare Contact Lens — Commercially available contact lens without a sensor
Device: Clinical IOP Measure — clinical IOP
  Other Names: iCare; Goldmann
Device: Experimental Contact Lens Sensor — Sensor contact lens being studied

SUMMARY:
This study is exploring the effectiveness and safety of soft contact lenses with embedded sensors, called smart contact lenses. Smart contact lenses are used to measure the pressure inside the eye.

DETAILED DESCRIPTION:
Subjects first present for a single qualification visit (phase 1), then present for up to 3 short-term (~1 hour) in-clinic visits (phase 2), and finally have visits prior to and following a full day (phase 3). Efficacy outcomes of the smart contact lens are compared to standard clinical measures of eye pressure. Safety outcomes of the smart contact lens are compared to those of traditional soft contact lenses.

ELIGIBILITY:
Glaucomatous Arm Inclusion Criteria

* 22+ years of age
* Able to wear soft contact lenses
* Previously diagnosed, currently pharmaceutically treated Primary Open Angle Glaucoma (POAG)

Non-Glaucomatous (Healthy Older Adults) Arm Inclusion Criteria

* 22+ years of age
* Able to wear soft contact lenses
* Without glaucomatous disease

Exclusion Criteria for all arms:

* Unable to complete the study procedures
* Ocular disease other than glaucoma (if applicable)
* Significant acute or chronic medical, neurologic, or other illness in the patient that, in the judgment of the Principal Investigator, could compromise subject safety, limit the ability to complete the study, and/or compromise the objectives of the study and/or is contradicted for soft contact lens or sensor lens use

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-19 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Goldmann Applanation Intraocular Pressure | Phase 2: 1 hour on 3 days Phase 3: Up to 14 hours on 3 days
  The IOP of participants will be measured with the Goldmann applanation tonometry (GAT) prior to and following device use, and in the contralateral eye during device use. A >2 mmHg difference in is considered clinically significantly different.
I-Care Tonometry Intraocular Pressure | Phase 2: 1 hour on 3 days Phase 3: Up to 14 hours on 3 days
  The I-Care (I-Care, Inc.) tonometry will also be evaluated during contralateral eye device use. A >2 mmHg difference in is considered clinically significantly different.
Lens comfort | Phase 2: 1 hour on 3 days Phase 3: Up to 14 hours on 3 days
  Participant-reported comfort will be assessed using a simple 100-point numeric scale where a rating of '100' represents extremely uncomfortable/intolerable and a rating of '1' perfectly comfortable/not noticeable at all. Comfort assessments will occur prior to, during, and following all device use to allow comparisons to typical or comparator devices. A 7-point difference in ratings is considered clinically significantly different.
Lens Fit | Phase 2: 1 hour on 3 days Phase 3: Up to 14 hours on 3 days
  Lens fit will be measured with slit lamp during lens wear and graded using the Cornea and Contact Lens Research Unit (CCLRU) grading scale, which ranges from 0 to 4 with a rating of 0 representing an optimal outcome. A difference of 1.0 grading unit will be considered clinically significant.

OTHER OUTCOMES:
Safety Outcome - Ocular Health | Phase 1: Day 1 Phase 2: Days 1, 2, and 3 Phase 3: Days 1, 2, and 3
  Investigator rated ocular health (hyperemia, conjunctival indentation, corneal staining) (0-4 Efron grading scale, where a rating of 0 represents an optimal outcome). Ocular health gradings following device wear will be compared pre-device use and post-device use and comparator bare soft contact lens use. A change in ocular health of 2 on the grading scale is considered clinically significant.
Safety Outcome - Visual Acuity | Phase 1: Day 1 Phase 2: Days 1, 2, and 3 Phase 3: Days 1, 2, and 3
  LogMAR visual acuity will be measured using ETDRS charts. A 0.2 change in visual acuity is considered a clinically significant change.
Safety Outcome - Octopus Kinetic Visual Field | Phase 1: Day 1
  Visual field extent (horizontal and vertical) will be measured with a kinetic visual field (e.g. Octopus Visual field). A 30% decrease in rate of visual field progression can be reliably projected to have a significant effect on health-related quality of life.
Safety Outcome - Corneal Thickness/Swelling | Phase 1: Day 1 Phase 2: Days 1, 2, and 3 Phase 3: Days 1, 2, and 3
  Corneal thickness/swelling will be measured using anterior segment ocular coherence tomography (OCT). Corneal swelling should be <8% following lens wear.

CONTACTS AND LOCATIONS:
Overall Officials: Pete S Kollbaum, Principal Investigator — Indiana University
Locations (1):
- Indiana University - Clinical Optics Research Lab, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: October 19, 2025 - September 20, 2028
Access Criteria: Study team members at Purdue University will be able to access all de-identified data collected during the study. This data will be shared via a secure electronic transfer.